CLINICAL TRIAL: NCT00468130
Title: Efficacy of Aripiprazole Versus Placebo in the Reduction of Aggressive and Aberrant Behavior in Autistic Children
Acronym: Abilify
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Principal Investigator, Sherie Novotny, M.D., Assistant Professor, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0220055441
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Autism
Keywords: Aggression; Irritability; Global autism severity
MeSH Terms: conditions — Autistic Disorder; Aggression | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aripiprazole (Experimental): Subjects in the experimental group will receive Aripiprazole
  Interventions: Drug: Aripiprazole
- Placebo (Placebo Comparator): Subjects in the control group will receive sugar pill
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Aripiprazole — Subjects under 40 kg will be started on 2.5mg per day of aripiprazole for the first week and increased to 5 mg at week 2. If clinically indicated (partial improvement with minimal or no side effects), the dosage will be increased each week by 2.5 mg until they reach a maximum of 10 mg at week 4. Medication will not be increased after week four but may be lowered in the case of adverse effects. Subjects over 40 kg will start at 5 mg and be increased to 10 mg at week 2. If clinically indicated, they will be increased each week by 5 mg until they reach a maximum of 20 mg at week 4. After week 4, the subject will remain on the same stable dose, unless the dose needs to be decreased due to adverse effects
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Placebos — Inactive tablet made to resemble active tablet
  Subjects under 40 kg will be started on 2.5mg per day of placebo for the first week and increased to 5 mg at week 2. If clinically indicated (partial improvement with minimal or no side effects), the dosage will be increased each week by 2.5 mg until they reach a maximum of 10 mg at week 4. Medication will not be increased after week four but may be lowered in the case of adverse effects. Subjects over 40 kg will start at 5 mg and be increased to 10 mg at week 2. If clinically indicated, they will be increased each week by 5 mg until they reach a maximum of 20 mg at week 4. After week 4, the subject will remain on the same stable dose, unless the dose needs to be decreased due to adverse effects
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Hypothesis: (1) Aripiprazole treatment will be superior to placebo in reducing aggression and irritability in autistic individuals as shown by reductions in the Aberrant Behavior Checklist-irritability subscale.

(2) Aripiprazole treatment will be superior to placebo in the acute treatment of global autism severity.

The purpose of this study is to examine the possible benefit of the medication Aripiprazole in autistic individuals.

DETAILED DESCRIPTION:
Aripiprazole is an atypical antipsychotic medication which is currently approved for the treatment of schizophrenia in adults. Multiple clinical trials in both children and adults have shown the effectiveness in the treatment of autism with medications like Aripiprazole. This study aims at assessing the effect of aripiprazole vs. placebo treatment on symptoms of irritability and aggression associated with autism, as well as the effect on the global severity of child and adolescent autistic disorder. Children or adolescent outpatients, with age ranges from 5-17, will be enrolled into an 8-week placebo controlled, double blind treatment study. During the 8 weeks, patients will be monitored by the treating psychiatrist. Study assessments will be administered at designated time points.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV, ADI-R criteria for autistic disorder.
* Age 5-17 years.
* Outpatients
* Parent or legal guardian willing to sign informed consent.

Exclusion Criteria:

* Subject has been diagnosed with a psychotic disorder (such as schizophrenia) or a mood disorder, including depression or bipolar disorder (manic depression).
* Subject has caused visible harm to him/herself.
* Subject has an active seizure disorder or epilepsy (seizures within the past year).
* Subject has an unstable medical illness, including heart disease.
* Subject has experienced brain injury.
* Subject has a history of diabetes.
* Subject reports significant improvement of autism symptoms and behaviors to current medication or other therapies.
* Subject has a history of prior treatment with Aripiprazole of 5 mg/day or higher for 6 weeks.
* Subject lives in a far away area and/or does not have regular access to transportation to the clinical facility.
* Subject is a pregnant female or unwilling to use acceptable contraception if sexually active.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2006-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherie L. Novotny, MD, Principal Investigator — Child and Adolescent Psychiatry, UMDNJ
Locations (1):
- Department of Child and Adolescent Psychiatry, University Behavioral Health Care Building, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
No plan at this time.

REFERENCES:
- [Background] Aman M, Smgh N, Stewart A, Field C. The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects.Am J Ment Defic, 1985a;89(5):485 491 Campbell M, et al, Neuroleptic related dyskinesias in autistic children: a prospective longitudinal study, J Am Acad Child Adolesc Psychiatry 1997; 36(6): 835 43. Fomboime E. The epidemiology of autism: a review. Psychological Medicine, 1999; 29:769 786. Guy W. ECDEU assessment manual for psychopharmacology. Revised. NTMH Publication DHEW Publ No (adm.) 76 388. Bethesda, MD: National Institute of Mental Health, 1976; 217 222. McDougle CJ, Holmes JP, Bronson MR, Anderson GM, Volkmar FR, Price LH, Cohen DJ. Risperidone treatment of children and adolescents with pervasive developmental disorders: a prospective open label study. J Am Acad Child Adolesc Psychiatry. 1997 May;36(5):685 93. Stahl SM. Dopamine system stabilizers, aripiprazole, and the next generation of antipsychotics, J Clin Psychiatry. 2001;62(l1).
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- See also: Official site of the Division of Child and Adolescent Psychiatry — http://ubhc.umdnj.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects in the control group will receive sugar pill
  Placebos: Inactive tablet made to resemble active tablet
  Subjects under 40 kg will be started on 2.5mg per day of placebo for the first week and increased to 5 mg at week 2. If clinically indicated (partial improvement with minimal or no side effects), the dosage will be increased each week by 2.5 mg until they reach a maximum of 10 mg at week 4. Medication will not be increased after week four but may be lowered in the case of adverse effects. Subjects over 40 kg will start at 5 mg and be increased to 10 mg at week 2. If clinically indicated, they will be increased each week by 5 mg until they reach a maximum of 20 mg at week 4. After week 4, the subject will remain on the same stable dose, unless the dose needs to be decreased due to adverse effects
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 7 | 6
Completed | 5 | 4
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 6 | 13
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.3 (2) | 12.6 (2) | 12.4 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression Improvement (CGI-AD)
Description: Clinical Global Impression Improvement (CGI)-AD (Guy, 1976). This is a standard rating scale with 7-point global severity and change scales which has been modified for Autistic Disorder. A rating of 2 is given when there is a substantial reduction in symptoms so that a treating clinician would be unlikely to change treatment. A rating of 1 is reserved for patients who become virtually symptom-free. A rating of 3 (minimally improved) on the CGI is defined as slight symptomatic improvement that is not deemed clinically significant. Administration time is approximately 2 minutes. Minimum is 1 and maximum is 5. A lower score indicates improvement, whereas a higher score indicates worsening.
Time Frame: Administered weekly, initial and week 8 reported
Population: Participants were children with autism who enrolled in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 7 | 6
score on a scale
  Initial CGI score | 3.83 (0.41) | 4.25 (1.25)
  Week 8 CGI score | 2.67 (1.21) | 4.25 (1.5)

2. Secondary Outcome: Aberrant Behavior Checklist
Description: Aberrant Behavior Checklist (ABC) (irritability section) (Aman et al, 1985). The Aberrant Behavior Checklist assesses drug and other treatment effects on mentally retarded individuals. It consists of a five-factor scale comprising 58 items. We will use the Irritability section to assess aggressive and agitated behavior. While the internal consistency, validity and test-retest reliability were reported to be very good, inter-rater reliability was moderate (Aman et al, 1985). The ABC will be filled out by an informant, and then reviewed by the psychiatrist. Administration time is approximately 10 minutes. Maximum is 36, minimum is 0, a lower score indicates improvement.
Time Frame: Administered biweekly, initial and week 8 reported
Population: Participants were children with autism who enrolled in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Aripiprazole: Participants in the clinical trial who were given aripiprazole
- Placebo: Participants in the clinical trial who were given placebo
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 7 | 6
score on a scale
  Initial, Irritability | 15.67 (11.65) | 8.00 (4.58)
  Week 8, Irritability | 6.83 (6.7) | 8.67 (10.69)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the period of the active study. Adverse events for each participant were collected during that participants enrollment in the study, initial contact through end of study, an average of 12 weeks for each participant.
Description: One subject withdrew due to a worsening of his depression after discontinuing his antidepressant medication, after being randomized.
Arm/Group | Aripiprazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 1/7 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=7) | Placebo (N=6)
Worsening of depression (Nervous system disorders) | 1 (1) | 0 (0) — Worsening of depression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes